CLINICAL TRIAL: NCT05627869
Title: Comparison of Effects of Transversus Thoracic Muscle Plane Block vs Pecto-intercostal Fascial Block on Postoperative Opioid Consumption in Patients Undergoing Open Cardiac Surgery: A Prospective Randomized Study
Brief Title: Effects of TTPB vs PIFB on Opioid Consumption in Patients After Cardiac Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mariana Soliman, Lecturer of anaesthesia, surgical intensive care and pain managment, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mariana AbdElsayed
Record Dates: First submitted 2022-11-01; First posted 2022-11-28 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Pain; Postoperative
Keywords: TTPB; PIFB
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus thoracic muscle plane block (Active Comparator): TTPB group will receive bilateral ultrasound-guided transversus thoracic muscle plane block using 20 ml of bupivacaine 0.25% for each side.
  Interventions: Procedure: Transversus thoracic plane block
- Pecto-intercostal fascial plane block (Active Comparator): PIFB group will receive bilateral ultrasound-guided Pecto-intercostal fascial plane block using 20 ml of bupivacaine 0.25% for each side.
  Interventions: Procedure: Pecto intercostal fascial block

INTERVENTIONS:
Procedure: Transversus thoracic plane block — TTPB group will receive bilateral ultrasound-guided transversus thoracic muscle plane block using 20 ml of bupivacaine 0.25% for each side.
  Other Names: sunnypivacaine
  Arms: Transversus thoracic muscle plane block
Procedure: Pecto intercostal fascial block — PIFB group will receive bilateral ultrasound-guided Pecto-intercostal fascial plane block using 20 ml of bupivacaine 0.25% for each side.
  Other Names: sunnypivacaine
  Arms: Pecto-intercostal fascial plane block

SUMMARY:
The objective of this study is to compare the effects of TTPB vs PIFB on postoperative opioid consumption in patients undergoing open cardiac surgery.

DETAILED DESCRIPTION:
Cardiac surgery performed through median sternotomy is associated with significant postoperative pain.Poststernotomy pain leads to decreased patient satisfaction, delirium, cardiovascular complications (hypertension, tachycardia, arrhythmias), hyperglycemia and respiratory complications (bronchial secretion stasis, atelectasis and pneumonia).High-dose opioids can provide good postoperative analgesia for patients undergoing heart surgery. However, opioids have some side effects.The advent of ultrasound-guided regional anaesthesia led to the development of fascial plane chest wall block as transthoracic plane block and pectointercostal fascial block.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years.
2. Patient scheduled to undergo elective on-pump cardiac surgery with sternotomy.
3. American Society of Anesthesiologists classification of physical status < IV.

Exclusion Criteria:

1. Emergency surgery.
2. Off-pump surgery.
3. Redo surgery.
4. Ejection fraction less than 35%.
5. Refusal of the patient.
6. Known hypersensitivity to LA.
7. Chronic opioid use or chronic pain patient.
8. Psychiatric problems or communication difficulties.
9. Liver insufficiency (defined as a serum bilirubin ≥ 34 μmol/l, albumin ≤ 35 g/dl, INR ≥ 1.7)
10. Renal insufficiency (defined as a glomerular filtration rate < 44 ml/min).
11. Obstructive sleep apnea syndrome.
12. Coexisting hematologic disorders.
13. Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be total morphine consumption | 24 hours
  Total morphine consumption within 24 hours according Visual Analogue Score (VAS) for sternal pain both during rest and with cough (ranging from 0 indicating no pain to 10 indicating extreme pain). A score ≤ 3 was considered acceptable for pain relief. Supplementary rescue analgesia was administered in the form of morphine IV 0.05 mg/kg (at VAS ≥ 4).

SECONDARY OUTCOMES:
The secondary outcomes will be the first analgesic request time | 24 hours
  Is the time to ask for the first postoperative analgesia (morphine), and will be calculated from extubation to patient reporting Visual Analogue Score (VAS) ≥ 4.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana A Mansour, Lecturer, Principal Investigator — Benisuef university hospital
Locations (1):
- Benisuef University Hospital, Benisuef, Egypt

IPD SHARING:
Plan to Share IPD: No
TITLE

REFERENCES:
- [Derived] Mansour MA, Mahmoud HE, Fakhry DM, Kassim DY. Comparison of the effects of transversus thoracic muscle plane block and pecto-intercostal fascial block on postoperative opioid consumption in patients undergoing open cardiac surgery: a prospective randomized study. BMC Anesthesiol. 2024 Feb 10;24(1):63. doi: 10.1186/s12871-024-02432-w. PMID 38341525